CLINICAL TRIAL: NCT03103607
Title: Evaluation of the Disappearance of Graves' Orbitopathy in the Long Term
Brief Title: Disappearance of Graves' Orbitopathy
Acronym: DISGO
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Ricercatore (Assistant Professor), University of Pisa
Other Study IDs: DISGO
Record Dates: First submitted 2017-03-27; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ophthalmological evaluation — exophthalmometry, evaluation of the Clinical Activity Score (CAS), assessment of diplopia, measurement of visual acuity, assessment of the corneal status; examination of the fundi
Diagnostic Test: Questionnaire — Patients were asked to fill a questionnaire on self-perception related to GO with the following questions: i) are your eyes identical to the way they were before GO appeared?; ii) are your eyes normal? iii) do you have any limitations in daily activities related to your eyes?; iv) do you have any limitations in social life related to your eyes?

SUMMARY:
There is a general belief among physicians involved with Graves' orbitopathy (GO) that this syndrome is somehow "chronic", namely that the patient's eyes do not return the way they were before GO appeared.

The general impression that comes from the available studies is that the eyes of GO patients do not return to normal even after a very long time since the disease appearance under the physician's point of view, although a discrete proportion of patients feel so. However, no studies are available in which the issue was examined with both objective criteria and self-assessment.

The present study design was to investigated the disappearance of GO, regardless to treatment, in all consecutive patients with a history of GO of at least 10 years who came for a follow-up visit to our GO clinic over a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All GO patients with a GO history of at least 10 years who came for a follow-up visit in our GO clinic over a period of 5 consecutive years

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with GO
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Disappearance of GO | up to 18 years
  Absence of objective signs and subjective symptoms of GO GO was considered disappeared when all the following criteria were fulfilled: objective criteria: i) exophthalmos ≤19 mm in men and ≤17 mm in women; ii) clinical activity score ≤1/7 points; iii) absence of diplopia; iv) normal visual acuity; v) normal corneal status; vi) no GO-related alterations of the fundi; subjective criteria (questionnaire): i) perception of both eyes identical to the way they were before GO appeared; ii) perception of both eyes as normal; iii) no eye-related limitation in daily activities; and iv) no eye-related limitations in social life.

SECONDARY OUTCOMES:
Objective disappearance of GO | up to 18 years
  Absence of objective signs GO GO was considered disappeared when all the following criteria were fulfilled: i) exophthalmos ≤19 mm in men and ≤17 mm in women; ii) clinical activity score ≤1/7 points; iii) absence of diplopia; iv) normal visual acuity; v) normal corneal status; vi) no GO-related alterations of the fundi
Subjective disappearance of GO | up to 18 years
  Absence of subjective symptoms of GO GO was considered disappeared when all the following criteria were fulfilled: i) perception of both eyes identical to the way they were before GO appeared; ii) perception of both eyes as normal; iii) no eye-related limitation in daily activities; and iv) no eye-related limitations in social life.

IPD SHARING:
Plan to Share IPD: No